CLINICAL TRIAL: NCT02465320
Title: A Muticenter, Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy and Safety of a Single-Dose of COL-1077 in Women Undergoing Transvaginal Pipelle-Directed Endometrial Biopsy
Brief Title: COL-1077 (Lidocaine Bioadhesive Gel, 10%) in Women Undergoing Transvaginal Pipelle-Directed Endometrial Biopsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Juniper Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: COL-1077-07
Record Dates: First submitted 2015-06-01; First posted 2015-06-08 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Endometrial Biopsy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- COL-1077 (Active Comparator): lidocaine bioadhesive gel, 10%
  Interventions: Drug: COL-1077
- Placebo (Placebo Comparator): placebo bioadhesive gel
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: COL-1077 — single dose of 150mg lidocaine (10%w/w) administered by intravaginal insertion
  Other Names: lidocaine bioadhesive gel, 10%
  Arms: COL-1077
Drug: Placebo — single dose of bioadhesive gel administered by intravaginal insertion
  Other Names: bioadhesive gel
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if COL-1077 (10% lidocaine vaginal bioadhesive gel) will be effective as an acute-use anesthetic and can decrease the pain intensity associated with gynecologic procedures using endometrial biopsy as a representative procedure.

DETAILED DESCRIPTION:
COL-1077 is to be self-administered by patients prior to an outpatient transvaginal pipelle-directed endometrial biopsy with tenaculum placement in otherwise healthy women requiring biopsy.

ELIGIBILITY:
Inclusion Criteria:

1. Female with an intact uterus, who is ≥ 40 and ≤ 75 years of age
2. For those women who are thought to be postmenopausal, postmenopausal will be defined as at least 6 months of confirmed amenorrhea with follicle stimulating hormone (FSH) levels of ≥ 40.0 mIU/mL
3. Scheduled to undergo a planned pipelle-directed endometrial biopsy with tenaculum placement
4. Able to intravaginally self-administer the study drug using the supplied drug applicator and plunger (eg, have adequate manual dexterity)
5. Willing and able to attend all study visits and complete the pain assessments
6. Willing to abstain from sexual intercourse 24 hours prior to completion of the endometrial biopsy and for 24 hours following the endometrial biopsy
7. Women of childbearing potential must use adequate birth control measures during the course of the study and for at least 7 days after completing study treatment.
8. Read, understood, and provided written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization

Exclusion Criteria:

1. Pelvic inflammatory disease (PID) within the past 3 months of the Screening Visit (Visit 1) or any ongoing vaginal infection requiring intravaginal treatment
2. Coagulation disorders
3. Experiencing daily baseline pelvic or chronic pain
4. Experiencing menstruation or anticipated menstrual cycle during the study period
5. Currently using an intrauterine device (IUD) or vaginal ring
6. Has active vaginal, vulvar or cervical lesions, or cervical or uterine carcinoma
7. Women who are pregnant or lactating.
8. Known history of hypersensitivity, allergies or intolerance to lidocaine or other amino amide-type local anesthetics
9. Known allergy or intolerance to aspirin or non-steroidal anti-inflammatories
10. Participation in any other investigational drug or device trial within 30 days prior to the Screening Visit (Visit 1)
11. Regular use of any concomitant medications that might confound efficacy and/or safety assessments
12. Chronic pain conditions that require regular (eg, daily) use of analgesic and/or anti-inflammatory medications
13. Use of Class 1 antiarrhythmic or a history of clinically significant cardiac arrhythmia as determined by the investigator
14. History of severe acute or chronic medical or psychiatric condition or laboratory abnormality that could increase the risk associated with trial participation or trial drug administration or could interfere with the interpretation of trial results
15. Evidence of current alcohol or drug abuse.

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2015-05; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Pain Intensity recorded on the 11-point Numerical Pain Rating Scale (NPRS) | at the time of endometrial biopsy

SECONDARY OUTCOMES:
Pain intensity (using 11-point NPRS) | at the time of tenaculum placement, at the time of insertion of the pipelle, 1 minute following tenaculum removal, 5, 15, 30 and 60 minutes & 2, 6, 8, & 24 hours post-endometrial biopsy
Time-Weighted Average Pain Intensity (TWAPI) | time of tenaculum placement until 2 hours post-endometrial biopsy
Sum Pain Intensity Difference (SPID) | time of tenaculum placement until 2 & 8 hours post-endometrial biopsy
Rescue medication usage | up to 24 hours post-endometrial biopsy
  For those who used rescue medication, time to first dose of rescue medication & total number of rescue doses used will be determined
Proportion of responders vs. non-responders to COL-1077. | up to 24 hours post-endometrial biopsy

OTHER OUTCOMES:
Patient subjective assessment of study drug at the end of the study | up to 48 hours post-endometrial biopsy
  Patients will be asked to rate the study drug they received for pain by answering the following question. "How would you rate the study drug you received for pain?" Responses are to be recorded as poor (1), fair (2), good (3), or excellent (4)
Maximum plasma concentration (Cmax) | 1 hour prior to biopsy (baseline), 30 and 60 minutes, 2, 6, 8 and 24 hours post-endometrial biopsy
Area under the plasma concentration time curve (AUC) from time 0 to time of last quantifiable concentration (AUC0-last) | 1 hour prior to biopsy (baseline), 30 and 60 minutes, 2, 6, 8 and 24 hours post-endometrial biopsy
Time to maximum concentration ( tmax) | 1 hour prior to biopsy (baseline), 30 and 60 minutes, 2, 6, 8 and 24 hours post-endometrial biopsy
Apparent clearance (CL/F) | 1 hour prior to biopsy (baseline), 30 and 60 minutes, 2, 6, 8 and 24 hours post-endometrial biopsy
Terminal elimination half-life (t1/2) | 1 hour prior to biopsy (baseline), 30 and 60 minutes, 2, 6, 8 and 24 hours post-endometrial biopsy
Incidence of adverse events and serious adverse events as a measure of Safety and tolerability of COL-1077 | up to 7 calendar days post-study completion
  Incidence of adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Bridget A Martell, MA, MD, Study Director — Juniper Pharmaceuticals, Inc.
Locations (23):
- United States (23):
  - Futura Research, Norwalk, California
  - Bluebird Clinical Trials, Colorado Springs, Colorado
  - Red Rocks OB/GYN, Lakewood, Colorado
  - South Florida Medical Research, Aventura, Florida
  - Axcess Medical Research, Loxahatchee Groves, Florida
  - South Florida Clinical Research Institute, Margate, Florida
  - New Age Medical Research Corporation, Miami, Florida
  - Ideal Clinical Research, North Miami Beach, Florida
  - WR Mount Vernon Clinical Research, LLC, Sandy Springs, Georgia
  - Rosemark Women Care Specialist, Idaho Falls, Idaho
  - Women's Clinic of Lincoln PC, Lincoln, Nebraska
  - Accent Clinical Trial, Las Vegas, Nevada
  - Lawrence OB-GYN Clinical Research, LLC, Lawrenceville, New Jersey
  - Albany Medical College, Albany, New York
  - New York Center for Women's Health Research, New York, New York
  - Carolina Womens Research Wellness Center, Durham, North Carolina
  - Unified Women's Clinical Research - Greensboro, Greensboro, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Hawthorne Medical Research Inc., Winston-Salem, North Carolina
  - Lyndhurt Clinical Research (Unified Women's Clinical Research), Winston-Salem, North Carolina
  - Clinical Trials of South Carolina, Charleston, South Carolina
  - Physicians Research Options, Draper, Utah
  - North Spokane Women's Health, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Undecided